CLINICAL TRIAL: NCT05097768
Title: Effectiveness of Oral Premedication on the Success Rate of Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis: A Prospective, Double-blind, Randomized Controlled Trial
Brief Title: Effectiveness of Premedication on the Success Rate of Inferior Alveolar Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alfarabi Colleges (Other)
Responsible Party: Principal Investigator, Amr Elnaghy, Associate Professor of Endodontics, Alfarabi Colleges
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-8/1
Record Dates: First submitted 2021-10-17; First posted 2021-10-28 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Dexamethasone; Ketorolac; Tablets; Meloxicam; Ibuprofen

STUDY DESIGN:
Intervention Model Description: The trial will include five study groups, each consists of 50 patients who exhibits symptomatic irreversible pulpitis of a mandibular first or second molar. The patients will receive identically appearing capsules containing either dexamethasone 0.5 mg, ketorolac 10 mg, meloxicam 7.5 mg, ibuprofen 600 mg, or placebo by mouth 60 minutes before the administration of an IANB. Endodontic access will begin 15 minutes after completion of the IANB. The IANB success is defined as no or mild pain (Heft Parker visual analog scale recordings) on pulpal access or instrumentation.
Who Masked: Participant, Investigator
Masking Description: To blind the experiment, each of the 50 patients in each group will be randomly allocated a code consists of 2 letters and one number. Only the random numbers identify the medications; thus, the patient and doctor are uninformed of which medication will be given to them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dexamethasone (Active Comparator): Before the inferior alveolar nerve block injection by 60 minutes, the patient will receive Dexamethasone 0.5 mg.
  Interventions: Drug: Dexamethasone 0.5mg
- Ketorolac (Active Comparator): Before the inferior alveolar nerve block injection by 60 minutes, the patient will receive ketorolac 10 mg.
  Interventions: Drug: Ketorolac 10 Mg Oral Tablet
- Meloxicam (Active Comparator): Before the inferior alveolar nerve block injection by 60 minutes, the patient will receive meloxicam 7.5 mg.
  Interventions: Drug: Meloxicam 7.5 mg
- Ibuprofen (Active Comparator): Before the inferior alveolar nerve block injection by 60 minutes, the patient will receive ibuprofen 600 mg.
  Interventions: Drug: Ibuprofen 600 mg
- Placebo (Placebo Comparator): Before the inferior alveolar nerve block injection by 60 minutes, the patient will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone 0.5mg — The patients will be randomly given the medication by mouth 60 min before administering IANB.
  Arms: Dexamethasone
Drug: Ketorolac 10 Mg Oral Tablet — The patients will be randomly given the medication by mouth 60 min before administering IANB.
  Arms: Ketorolac
Drug: Meloxicam 7.5 mg — The patients will be randomly given the medication by mouth 60 min before administering IANB.
  Arms: Meloxicam
Drug: Ibuprofen 600 mg — The patients will be randomly given the medication by mouth 60 min before administering IANB.
  Arms: Ibuprofen
Drug: Placebo — The patients will be randomly given the medication by mouth 60 min before administering IANB.
  Arms: Placebo

SUMMARY:
Purpose: The aim of this prospective, double-blind, randomized controlled trial is to compare the effect of oral premedication of dexamethasone, ketorolac, meloxicam, ibuprofen or placebo on the success of inferior alveolar nerve blocks (IANB) of mandibular posterior teeth in patients experiencing symptomatic irreversible pulpitis. Methods: The trial will include five study groups, each consists of 50 patients who exhibits symptomatic irreversible pulpitis of a mandibular first or second molar. The patients will receive identically appearing capsules containing either dexamethasone 0.5 mg, ketorolac 10 mg, meloxicam 7.5 mg, ibuprofen 600 mg, or placebo by mouth 60 minutes before the administration of an IANB. Endodontic access will begin 15 minutes after completion of the IANB. The IANB success is defined as no or mild pain (Heft Parker visual analog scale recordings) on pulpal access or instrumentation.

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, placebo-controlled trial. This trial follows the most recent update of the Declaration of Helsinki criteria (October 2013). The Vision Colleges Research Ethics Committee approved the clinical trial protocol and informed consent. The Consolidated Standards of Reporting Trials guidelines will be used to report the present superiority study. Participants under the age of 18, those with a history of major medical issues, those who had used central nervous system depressants or any analgesic drug in the preceding 6 h, those who were pregnant, and those who were unable to give informed consent will be excluded from the study. All the patients will sign a consent form that had been approved.

The inclusion criteria will be active pain in the first or second mandibular molar, a prolonged response to cold testing, no periapical radiolucency on periapical radiographs, and a vital coronal pulp on access opening. The Modified Dental Anxiety Scale will be used to assess the patients' anxiety levels. The pain of the patients will be categorized into four categories using the Heft-Parker visual analogue scale (HP VAS):

0 mm: no pain 0-54 mm: faint, weak, or mild 55-114 mm: moderate pain >114 mm: strong, intense, and maximum possible Permuted block randomization will be used to ensure the homogeneity of the five groups. The patients will be randomly given dexamethasone 0.5 mg, ketorolac 10 mg, meloxicam 7.5 mg, ibuprofen 600 mg, or placebo by mouth 60 mins before administering IANB. To blind the experiment, each of the 50 patients in each group will be randomly allocated a code consists of 2 letters and one number. Only the random codes will identify the medications; thus, the patient and clinicians are uninformed of which medication will be given to them. At 60 mins after taking the medication or placebo, the operator will use a cotton tip applicator to put anaesthetic gel at the IANB injection site for 60 s.

The participants will then give regular IANB injections and 0.9 mL long buccal injections containing 2% lidocaine and 1:100,000 epinephrine. Each patient will be asked for lip numbness every 5 mins for 15 mins after the IANB. The block will be considered missed if substantial lip numbness was not reported by 15 mins, and the participant will be excluded from the trial. After the lip numbness is determined, the tooth will be isolated and a second cold test will be performed to verify the presence or absence of any painful reaction.

After that, the endodontic access will be conducted. During the endodontic process, patients will be asked to rate any pain they experienced. If the patient is in pain, the treatment will be stopped, and the patient will use the HP VAS to rate his/her discomfort. The success of the IANB is identified by the capability to access and clean and shape the root canal space without pain (VAS score of 0) or mild pain (VAS rating ≤54 mm). The rubber dam will be removed if the patient had moderate or severe pain (VAS rating ≥ 55 mm). Then, a buccal infiltration of a cartridge containing 4% articaine with 1:100,000 epinephrine will be given buccally to the tooth that required emergency treatment. After 5 mins, the rubber dam will be replaced, and endodontic access will be resumed. The capability to access and instrument the tooth without pain (VAS score of 0) or with mild pain (VAS rating ≤54 mm) is considered a success of the buccal infiltration. Intraosseous anesthesia will be given to the patients who still had moderate to severe pain. The intraosseous injection will be given. If that didn't work, an intrapulpal injection will be given, followed by endodontic debridement. The extent of access preparation and/or instrumentation will be recorded as within dentine, within pulp space, and instrumentation of canals.

The VAS satisfaction form will be used to record the post-treatment satisfaction of the patient. On the VAS (0-100 mm), the patient will be asked to draw a vertical line to represent their experience with the entire treatment. The VAS is classified into four categories; 0: not satisfied, >0 mm and ≤33 mm: somewhat satisfied, >33 mm but <66 mm: moderately satisfied and ≥66 mm: completely satisfied.

ELIGIBILITY:
Inclusion Criteria:

* active pain in a mandibular molar first or/and the second molar
* prolonged response to cold testing
* absence of any periapical radiolucency on periapical radiographs
* vital coronal pulp on access opening
* able to give informed consent

Exclusion Criteria:

* less than 18 years old
* history of serious medical problems
* used central nervous system depressants or any analgesic medication within the previous 6 hours
* pregnancy
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Pain Measurement as it will be assessed on a Heft-Parker 170 mm Visual Analog Scale | 15 minutes after the inferior alveolar nerve block
  At 60 minutes after receiving the medication or placebo, the participants will be given inferior alveolar nerve block injection. Each patient will be asked for lip numbness every 5 minutes for 15 minutes after inferior alveolar nerve block injection. During the endodontic process, patients will be asked to rate any pain they experienced on a Heft-Parker visual analog scale. The number of millimeters along the scale will be reported. No pain corresponded to 0 mm. Mild pain is defined as greater than 0 mm and less than or equal to 54 mm. Mild pain is the descriptors of "faint", "weak", and "mild pain". Moderate pain is defined as greater than 54 mm and less than 114 mm and includes the descriptor "moderate". Severe pain is defined as equal to or greater than 114 mm up to and including 170 mm. Severe pain includes the descriptors of "strong", "intense", and "maximum possible."

SECONDARY OUTCOMES:
Postoperative Satisfaction on a 100 mm Visual Analog Scale | Immediately post-procedure on Day 0
  Patients will rate their level of satisfaction after treatment procedure using a visual analog scale. The scale ranges from "not satisfied," to "somewhat satisfied," to "moderately satisfied," to "completely satisfied." Not satisfied corresponded to 0 mm. Somewhat satisfied is defined as greater than 0 mm and less than or equal to 33 mm. Moderately satisfied is defined as greater than 33 mm and less than 66 mm. Completely satisfied is defined as equal to or greater than 66 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Elnaghy, PhD, Principal Investigator — Vision Colleges
Locations (1):
- Vission Colleges, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagendrababu V, Pulikkotil SJ, Veettil SK, Teerawattanapong N, Setzer FC. Effect of Nonsteroidal Anti-inflammatory Drug as an Oral Premedication on the Anesthetic Success of Inferior Alveolar Nerve Block in Treatment of Irreversible Pulpitis: A Systematic Review with Meta-analysis and Trial Sequential Analysis. J Endod. 2018 Jun;44(6):914-922.e2. doi: 10.1016/j.joen.2018.02.017. Epub 2018 Apr 27. PMID 29709297
- [Background] Pulikkotil SJ, Nagendrababu V, Veettil SK, Jinatongthai P, Setzer FC. Effect of oral premedication on the anaesthetic efficacy of inferior alveolar nerve block in patients with irreversible pulpitis - A systematic review and network meta-analysis of randomized controlled trials. Int Endod J. 2018 Sep;51(9):989-1004. doi: 10.1111/iej.12912. Epub 2018 Mar 24. PMID 29480930
- [Background] Yadav M, Grewal MS, Grewal S, Deshwal P. Comparison of Preoperative Oral Ketorolac on Anesthetic Efficacy of Inferior Alveolar Nerve Block and Buccal and Lingual Infiltration with Articaine and Lidocaine in Patients with Irreversible Pulpitis: A Prospective, Randomized, Controlled, Double-blind Study. J Endod. 2015 Nov;41(11):1773-7. doi: 10.1016/j.joen.2015.06.008. Epub 2015 Sep 26. PMID 26410153
- [Background] Aggarwal V, Singla M, Kabi D. Comparative evaluation of effect of preoperative oral medication of ibuprofen and ketorolac on anesthetic efficacy of inferior alveolar nerve block with lidocaine in patients with irreversible pulpitis: a prospective, double-blind, randomized clinical trial. J Endod. 2010 Mar;36(3):375-8. doi: 10.1016/j.joen.2009.11.010. PMID 20171350